CLINICAL TRIAL: NCT02044159
Title: Steroid Use in Pediatric Fluid and Vasoactive Infusion Dependent Shock - Pilot Study (STRIPES)
Brief Title: Steroid Use in Pediatric Fluid and Vasoactive Infusion Dependent Shock - Pilot Study
Acronym: STRIPES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Alberta Children's Hospital (Other); British Columbia Children's Hospital (Other); London Health Sciences Centre (Other); St. Justine's Hospital (Other); IWK Health Centre (Other); Montreal Children's Hospital of the MUHC (Other)
Responsible Party: Principal Investigator, Kusum Menon, Senior Investigator, CHEO Research Institute; Associate Professor, University of Ottawa; Physician, Division of Critical Care, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STRIPES-Pilot
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Shock
Keywords: Hydrocortisone; Pediatrics; Adrenal Insufficiency
MeSH Terms: conditions — Shock; Adrenal Insufficiency | interventions — Hydrocortisone; hydrocortisone hemisuccinate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrocortisone (Experimental): Patients randomized to the hydrocortisone arm will receive a 2 mg/kg hydrocortisone IV bolus on enrolment followed by 1 mg/kg of hydrocortisone IV q6h until the patient has not had an escalation in therapy for at least 12 hours. If the patient meets these criteria their hydrocortisone will be weaned to 1 mg/kg every 8 hours which will be continued until they are off all vasoactive infusions for 12 hours. If following the initial hydrocortisone wean, the patient requires fluid boluses and/or an increase in their vasoactive infusion(s), their hydrocortisone will be increased back to 1 mg/kg of hydrocortisone IV q6h until they meet stability criteria again. Duration of treatment will range from a minimum of 20 hours to a maximum of 7 days of study drug.
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator): Patients randomized to the placebo arm will receive a placebo solution consisting of normal saline equivalent in volume to the appropriate dose of hydrocortisone. Hydrocortisone and placebo will be identical in appearance, volume and smell as hydrocortisone is made up in normal saline and dissolves completely with no visible precipitate. The dosing regimen will be identical to the hydrocortisone arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone will be made up as a 10 mg/ml solution so the volume of added fluid will be very small (2 to 10 mls even for the initial dose of 2 mg/kg).
  Other Names: SOLU-CORTEF
  Arms: Hydrocortisone
Other: Placebo — The placebo (normal saline) will be identical in appearance, volume and smell to the active study drug (hydrocortisone).
  Other Names: Placebo (saline solution)
  Arms: Placebo

SUMMARY:
Approximately 20,000 children per year in North America present to the hospital with severe shock. Children who develop this condition have very low blood pressures and as a result may suffer damage to their internal organs and may even die. Some children with this condition may significantly benefit from the use of steroids but steroids in such patients may also have potential side effects. Therefore it is important to study the use of steroids carefully in these children. The STRIPES research program will examine the effectiveness and safety of steroids in children. Before conducting a large, randomized controlled trial (RCT), a pilot study (STRIPES Pilot Study) will be conducted in multiple sites across Canada. The STRIPES Pilot Study will allow testing of the STRIPES study protocol in a smaller group of patients.

DETAILED DESCRIPTION:
This study is a multi-centre pilot RCT to determine the feasibility of doing a full trial on the effect of steroids versus placebo in children with fluid and vasoactive infusion dependent shock. The principal investigator and colleagues recently published two articles on this topic which were selected as the Feature Article and Feature Review in the June edition of Pediatric Critical Care Medicine. Both of these publications strongly support the interest in this area and the accompanying editorial strongly supported the need for a well-designed RCT.

RATIONALE: Approximately 20,000 children per year present to emergency departments, pediatric wards and intensive care units in North America with fluid and vasoactive infusion dependent shock. This severe type of shock results in significant morbidity and carries a 2-10% mortality rate depending on the setting in which it occurs. This form of shock is thought to arise from dysfunction of the hypothalamic-pituitary-adrenal axis through a variety of mechanisms and has been referred to as relative adrenal insufficiency or critical illness related adrenal insufficiency. Many clinicians believe that corticosteroids improve outcomes in such patients and therefore use them when confronted with a critically ill child with fluid and vasoactive infusion dependent shock. However, the effectiveness and safety of steroid replacement therapy in pediatric shock remain to be demonstrated.

OBJECTIVES - PILOT STUDY: Before embarking on a multi-centre definitive trial to address the questions listed above, the STRIPES Pilot Study has 3 specific feasibility objectives: 1) To estimate the rate of patient recruitment and understand barriers to recruitment; 2) To assess adherence to our specific treatment protocol; and 3) To document the frequency of and understand the reasons for open label steroid use.

OBJECTIVES - FULL RCT: Following successful completion of the STRIPES Pilot Study, the next phase will be a large, multi centre RCT to answer the following questions: 1) What is the effect of hydrocortisone versus placebo on the time to discontinuation of vasoactive agents among pediatric patients with fluid and vasoactive infusion dependent shock?; and 2) In patients with fluid and vasoactive infusion dependent shock, what is the effect of hydrocortisone versus placebo on i) pediatric intensive care unit (PICU) mortality; ii) duration of mechanical ventilation; iii) new onset of organ dysfunction; iv) PICU length of stay; and v) incidence of adverse events?

RESEARCH PLAN: The STRIPES Pilot Study is designed as a pragmatic, multi-centre, double blind, RCT of intravenous hydrocortisone versus intravenous placebo in fluid and vasoactive infusion dependent shock. This study aims to enroll 72 patients from 7 pediatric centres across Canada over a one year period. Patients will be recruited from the Emergency Department and the PICU within 6 hours of being stared on a vasoactive agent. Research ethics board approval will be obtained from all participating centres and application for deferred consent will be made at 5 sites. Health Canada approval is not required as hydrocortisone is approved for use in children at the doses and for the indication for which it is being used in this study.

As part of the pragmatic design, the prescriptive component of the protocol will be limited to the administration and weaning of the study drug. The requirement for intubation, mechanical ventilation, sedation and analgesia, use of hemodynamic triggers and endpoints, red cell transfusions, antibiotics and fluid boluses will be left to the discretion of the treating physician. The Surviving Sepsis Guidelines Flowchart will be attached to the study protocol for easy reference by the treating physician but its use will not be mandated; however, the use of vasoactive infusions and other therapies will be recorded. The proposed duration of treatment will range from a minimum of 20 hours to a maximum of 7 days of study drug. Outcome data, including survival status and frequency of adverse events, will be collected daily until discharge from hospital.

Although the primary focus of this pilot study is to determine the feasibility of conducting a clinical outcome based RCT of steroids versus placebo in shock, this pilot also provides an excellent opportunity to perform some exploratory mechanistic studies. These will include 1) comparison of total and free cortisol levels of patients with shock; 2) measurement of stratification biomarkers; and 3) determination of 25 hydroxyvitamin D and 1,25 hydroxyvitamin D levels on admission. Patients with access for blood sampling and for whom consent has been obtained will have blood samples sent for these mechanistic studies.

Patients will be randomized to the hydrocortisone or placebo arm using web-based, centralized permuted block randomization, stratified by centre. All study personnel (the overall study research coordinator, research assistants, site investigators, principal investigator, co-investigators, data management personnel, and statisticians), members of the health care team (treating physicians, bedside nurses, and clinical pharmacists) and patients/families will be blinded to the study group assignment.

SIGNIFICANCE: Results of the STRIPES Pilot Study will provide essential feasibility data for planning and conducting a larger, multi-centre trial that will help to establish the role of steroids in children with fluid and vasoactive infusion dependent shock. There are special challenges to patient recruitment in critically ill pediatric populations, adherence to treatment protocols and to the limitation of open label use of steroids, all of which the STRIPES Pilot study will help to address. Success of the STRIPES Pilot Study will be based on the ability to achieve each of the three feasibility objectives listed above. If the pilot study demonstrates feasibility, no major protocol changes are needed, and no safety concerns are raised by the Data Safety Monitoring Board, then the results of the pilot study will be rolled into the full trial. However, if any of the above criteria are not met, then the protocol will be re-evaluated and the feasibility results of the pilot study published independently.

ELIGIBILITY:
Inclusion Criteria:

* Children newborn to 17 years
* On any dose of any vasoactive infusion for between 1 to 6 hours

Exclusion Criteria:

* Patients who have known or suspected hypothalamic, pituitary or adrenal disease
* Patients who are currently receiving steroids for the treatment of shock/suspected shock prior to randomization
* Patients who are expected to have treatment withdrawn
* Patients who are premature infants (<38 weeks corrected gestational age)
* Patients who are pregnant
* Patients post cardiac surgery
* Patient who received their first dose of vasoactive infusion >24 hours after PICU admission
* Patient who is no longer on vasoactive infusion at the time of study enrollment, and/or is expected to no longer be on vasoactive infusion at the time the first dose of study drug will be administered
* Patients for whom primary cardiogenic shock is strongly suspected
* Patients for whom spinal shock is strongly suspected
* Patients for whom hemorrhagic or hypovolemic shock is strongly suspected
* Patients who were previously enrolled in the STRIPES study
* Patients who receive a vasoactive agent for reasons not related to shock
* Physician refusal

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kusum Menon, MD, MSc, Principal Investigator — Children's Hospital of Eastern Ontario; Karen Choong, MB, MSc, Study Chair — McMaster Children's Hospital; James D McNally, MD, PhD, Study Chair — Children's Hospital of Eastern Ontario; Lauralyn McIntyre, MD, MSc, Study Chair — The Ottawa Hospital; Margaret Lawson, MD, MSc, Study Chair — Children's Hospital of Eastern Ontario; Hector Wong, MD, Study Chair — Children's Hospital Medical Center, Cincinnati; Tim Ramsay, MSc, PhD, Study Chair — Ottawa Hospital Research Institute
Locations (7):
- Canada (7):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Hospital St. Justine, Montreal, Quebec

REFERENCES:
- [Background] Menon K, McNally JD, Choong K, Ward RE, Lawson ML, Ramsay T, Wong HR. A survey of stated physician practices and beliefs on the use of steroids in pediatric fluid and/or vasoactive infusion-dependent shock. Pediatr Crit Care Med. 2013 Jun;14(5):462-6. doi: 10.1097/PCC.0b013e31828a7287. PMID 23628832
- [Background] Menon K, McNally D, Choong K, Sampson M. A systematic review and meta-analysis on the effect of steroids in pediatric shock. Pediatr Crit Care Med. 2013 Jun;14(5):474-80. doi: 10.1097/PCC.0b013e31828a8125. PMID 23867428
- [Background] Odetola FO, Gebremariam A, Freed GL. Patient and hospital correlates of clinical outcomes and resource utilization in severe pediatric sepsis. Pediatrics. 2007 Mar;119(3):487-94. doi: 10.1542/peds.2006-2353. PMID 17332201
- [Background] Kissoon N, Carcillo JA, Espinosa V, Argent A, Devictor D, Madden M, Singhi S, van der Voort E, Latour J; Global Sepsis Initiative Vanguard Center Contributors. World Federation of Pediatric Intensive Care and Critical Care Societies: Global Sepsis Initiative. Pediatr Crit Care Med. 2011 Sep;12(5):494-503. doi: 10.1097/PCC.0b013e318207096c. PMID 21897156
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Menon K, Ward RE, Lawson ML, Gaboury I, Hutchison JS, Hebert PC; Canadian Critical Care Trials Group. A prospective multicenter study of adrenal function in critically ill children. Am J Respir Crit Care Med. 2010 Jul 15;182(2):246-51. doi: 10.1164/rccm.200911-1738OC. Epub 2010 Mar 18. PMID 20299532
- [Background] Zimmerman JJ, Barker RM, Jack R. Initial observations regarding free cortisol quantification logistics among critically ill children. Intensive Care Med. 2010 Nov;36(11):1914-22. doi: 10.1007/s00134-010-2007-1. Epub 2010 Aug 19. PMID 20721535
- [Background] Poomthavorn P, Lertbunrian R, Preutthipan A, Sriphrapradang A, Khlairit P, Mahachoklertwattana P. Serum free cortisol index, free cortisol, and total cortisol in critically ill children. Intensive Care Med. 2009 Jul;35(7):1281-5. doi: 10.1007/s00134-009-1480-x. Epub 2009 Apr 8. PMID 19352620
- [Background] Hamrahian AH, Oseni TS, Arafah BM. Measurements of serum free cortisol in critically ill patients. N Engl J Med. 2004 Apr 15;350(16):1629-38. doi: 10.1056/NEJMoa020266. PMID 15084695
- [Background] Pollack MM, Patel KM, Ruttimann UE. PRISM III: an updated Pediatric Risk of Mortality score. Crit Care Med. 1996 May;24(5):743-52. doi: 10.1097/00003246-199605000-00004. PMID 8706448
- [Background] Zimmerman JJ, Donaldson A, Barker RM, Meert KL, Harrison R, Carcillo JA, Anand KJ, Newth CJ, Berger J, Willson DF, Jack R, Nicholson C, Dean JM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Real-time free cortisol quantification among critically ill children. Pediatr Crit Care Med. 2011 Sep;12(5):525-31. doi: 10.1097/PCC.0b013e3181fe4474. PMID 21057361
- [Background] Boonen E, Vervenne H, Meersseman P, Andrew R, Mortier L, Declercq PE, Vanwijngaerden YM, Spriet I, Wouters PJ, Vander Perre S, Langouche L, Vanhorebeek I, Walker BR, Van den Berghe G. Reduced cortisol metabolism during critical illness. N Engl J Med. 2013 Apr 18;368(16):1477-88. doi: 10.1056/NEJMoa1214969. Epub 2013 Mar 19. PMID 23506003
- [Background] Watson RS, Carcillo JA, Linde-Zwirble WT, Clermont G, Lidicker J, Angus DC. The epidemiology of severe sepsis in children in the United States. Am J Respir Crit Care Med. 2003 Mar 1;167(5):695-701. doi: 10.1164/rccm.200207-682OC. Epub 2002 Nov 14. PMID 12433670
- [Background] Wong HR, Cvijanovich NZ, Allen GL, Thomas NJ, Freishtat RJ, Anas N, Meyer K, Checchia PA, Lin R, Shanley TP, Bigham MT, Wheeler DS, Doughty LA, Tegtmeyer K, Poynter SE, Kaplan JM, Chima RS, Stalets E, Basu RK, Varisco BM, Barr FE. Validation of a gene expression-based subclassification strategy for pediatric septic shock. Crit Care Med. 2011 Nov;39(11):2511-7. doi: 10.1097/CCM.0b013e3182257675. PMID 21705885
- [Background] McNally JD, Doherty DR, Lawson ML, Al-Dirbashi OY, Chakraborty P, Ramsay T, Menon K. The relationship between vitamin D status and adrenal insufficiency in critically ill children. J Clin Endocrinol Metab. 2013 May;98(5):E877-81. doi: 10.1210/jc.2013-1126. Epub 2013 Apr 1. PMID 23547046
- [Derived] O'Hearn K, McNally D, Choong K, Acharya A, Wong HR, Lawson M, Ramsay T, McIntyre L, Gilfoyle E, Tucci M, Wensley D, Gottesman R, Morrison G, Menon K; Canadian Critical Care Trials Group. Steroids in fluid and/or vasoactive infusion dependent pediatric shock: study protocol for a randomized controlled trial. Trials. 2016 May 6;17(1):238. doi: 10.1186/s13063-016-1365-6. PMID 27153945

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrocortisone | Placebo
Started (Fifty-seven patients were randomized (86.4%, 57/66 approached for consent)) | 27 | 30
Completed | 23 | 26
Not Completed | 4 | 4
Not completed — Consent declined (deferred consent) | 2 | 4
Not completed — No longer eligible, drug not given | 1 | 0
Not completed — Nurse declined to give study drug | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocortisone | Placebo | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 90.0 [14.3 to 155.8] | 108.0 [44.5 to 146.5] | 92.0 [37.5 to 150.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 12 | 13 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patient Accrual Rate Over One Year (% of Target Sample Size Achieved)
Description: The total number of participants recruited over the recruitment period to both arms (this was a feasibility outcome that was analyzed for the full cohort and, as stated a priori in the study protocol was not compared between study arms). Our goal is to recruit 72 patients over one year . However, we will consider patient accrual rate to be adequate if we recruit 60 patients from seven sites within this time period.
Time Frame: 1 year
Population: This feasibility objective, as stated a priori in the protocol, was analyzed for the full study cohort and was not compared between arms. The primary objective was the patient accrual rate over one year (percentage of for the target sample size for the full cohort that was achieved).
Measure: Number; unit: percentage of target sample size
Groups:
- Full Cohort: Feasibility outcomes were analyzed for the full cohort, and not compared between groups
Arm/Group | Full Cohort
Number analyzed (Participants) | 57
percentage of target sample size | 82

2. Secondary Outcome: 1a. Time to Administration of the First Dose of Study Drug
Description: This objective is a measure of protocol adherence. The goal is to have patients randomized within 6 hours, and study drug administration completed within 8 hours of starting a vasoactive medication. We will consider adherence to our protocol to be adequate if secondary outcomes 1a to 1c are met in 80% of enrolled patients.
Time Frame: 8 hours from starting vasoactive medication
Population: This feasibility objective, as stated a priori in the protocol, was analyzed for the full study cohort and was not compared between arms. Objective 1a was to determine the time to administration of the first dose of study drug for the full cohort.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Full Cohort: Feasibility objectives were assessed for the full cohort, and not compared between study arms
Arm/Group | Full Cohort
Number analyzed (Participants) | 49
hours | 3.8 (2.6)

3. Secondary Outcome: 1b. Weaning of Study Drug to q8h When Patient is Hemodynamically Stable
Description: This objective is a measure of protocol adherence. The goal is weaning of study drug to q8h within 12 hours of no escalation of therapy. We will consider adherence to our protocol to be adequate if secondary outcomes 1a to 1c are met in 80% of enrolled patients.
Time Frame: 7 days
Population: The percentage of study drug doses administered correctly was calculated for the full cohort.This feasibility objective was analyzed for the full cohort, and as stated a prior in our protocol, was not compared between study arms.
Measure: Number; unit: % of doses administered correctly
Arm/Group | Full Cohort
Number analyzed (Participants) | 49
% of doses administered correctly | 97.6

4. Secondary Outcome: 1c. Discontinuation of Study Drug When Off All Vasoactive Medications
Description: This objective is a measure of protocol adherence. The goal is to discontinue study drug within 12 to 18 hours of vasoactive medications being stopped. We will consider adherence to the protocol adequate if secondary outcomes 1a to 1c are met in 80% of enrolled patients.
Time Frame: 7 days
Population: The percentage of study drug doses that were administered correctly for the full cohort.This feasibility objective, as stated a priori in the protocol, was analyzed for the full study cohort and was not compared between arms.
Measure: Number; unit: % of doses administered correctly
Arm/Group | Full Cohort
Number analyzed (Participants) | 49
% of doses administered correctly | 97.6

5. Secondary Outcome: Number of Patients Started on Open Label Steroids by the Treating Physician
Description: We will consider the number of patients started on open label steroids by the treating physician to be acceptable if it occurs in less than 10% of patients. We will also collect information on the clinical parameters of patients when open label steroids are given.
Time Frame: 7 days
Population: The total number (and %) of patients in the full cohort who were administered open-label steroids by the treating physician.This feasibility objective, as stated a priori in the protocol, was not compared or reported separately by study arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Cohort
Number analyzed (Participants) | 49
Participants | 6

6. Secondary Outcome: Time to Discontinuation of Vasoactive Infusions
Description: The time to discontinuation of vasoactive agents will be used to better estimate the sample size for the full study.
Time Frame: Daily during hospital admission (up to 28 days)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 23 | 26
hours | 38.2 [13.2 to 71.3] | 33.1 [19.4 to 59.1]

7. Secondary Outcome: Number of Participants With Incidence of Adverse Events and Mortality in the Full Cohort
Description: The specific adverse events that will be measured include: severe bleeding, secondary infections and the use of insulin infusions. The incidence of adverse events and mortality rate was measured in aggregate (i.e. the whole cohort) in order to provide a better baseline estimate of these outcomes in our study population.
Time Frame: Daily during hospital admission (up to 28 days)
Population: The number of participants with incidence of adverse events and mortality rate in the full cohort in order to provide a better baseline estimate of these outcomes in our study population.
Measure: Count of Participants; unit: Participants
Groups:
- Full Cohort: Measured in aggregate for full cohort
Arm/Group | Full Cohort
Number analyzed (Participants) | 49
Participants | 24

8. Secondary Outcome: Percentage of Patients for Whom Blood Samples Are Sent, and Successfully Received and Analyzed in Their Respective Labs
Description: A total of 3 ml of blood in a red top tube will be collected within 24 hours of hospital admission. Patients with access for blood sampling and for whom consent has been obtained will have blood samples collected. The samples will be separated at each centre, stored until the end of the recruitment period, and then shipped to the principal investigators's centre as per the specific test requirements. The free cortisol and stratification biomarker samples will be batched and then shipped to Cincinnati for analysis at the end of the study. The number of samples collected, and the number of samples successfully received and analyzed at the principal investigator's site and at the Cincinnati lab will be determined at the end of the recruitment phase.
Time Frame: End of the study recruitment phase (up to 1.5 years)
Population: The total number of patients in the full cohort for whom a study blod sample was collected, received and analyzed. This feasibility outcome, as stated a priori in the study protocol, was analyzed for the full cohort and was not compared between arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Cohort
Number analyzed (Participants) | 49
Participants | 44

ADVERSE EVENTS:
Arm/Group | Hydrocortisone | Placebo
All-Cause Mortality (participants affected / at risk) | 1/23 | 3/26
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 12/23 | 8/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone (N=23) | Placebo (N=26)
Gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2) | 2 (2)
New infection (Infections and infestations) | 6 (6) | 5 (5)
Insulin infusion (Endocrine disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No